CLINICAL TRIAL: NCT00242658
Title: Computerized Physical Activity Promotion in Primary Care
Brief Title: Computerized Health Education to Promote Physical Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 269; 7R01HL067005-03 (NIH); 02F.214 CHIP; NCT00201032 (obsolete NCT alias)
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension
Keywords: Physical Activity; Wellness Programs; Health Promotion; Blood Pressure, High
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Physical Activity Intervention Group (Experimental): Four feedback reports aimed to increase physical activity.
  Interventions: Behavioral: Tailored Physical Activity Intervention
- No Tailored Physical Activity Intervention Group (No Intervention): General reports on preventive screening based on responses to preventive screening questions.

INTERVENTIONS:
Behavioral: Tailored Physical Activity Intervention — Tailored physical activity computer reports will be provided to patients and physicians.
  Other Names: Exercise Intervention
  Arms: Tailored Physical Activity Intervention Group

SUMMARY:
This study will test the efficacy of providing primary care physicians and their patients with computer-tailored information, based on patients' responses to survey questions. The health education messages are designed to encourage patients to become physically active and to encourage physicians to counsel their patients about exercise.

DETAILED DESCRIPTION:
The main objective of this study is to determine, via a 6-month randomized controlled study, the efficacy of providing tailored physical activity computer reports to patients and physicians. The primary outcome is minutes of physical activity measured by the 7-Day Physical Activity Recall interview at 6 months. The intervention group completed physical activity surveys at baseline, 1, 3, and 6 months. Based on their responses, participants received four feedback reports at each time point. The reports aimed to motivate participants to increase physical activity, personalized to participants' needs; they also included an activity prescription. The control group received identical procedures, except that they received general reports on preventive screening based on their responses to preventive screening questions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and read English
* Current patient of a physician participating in this study (if selecting a new physician, may deliberately select one that is involved in the study, in order to participate)
* Ability to complete all written surveys
* Accessible for follow-up telephone surveys
* Ability to undergo exercise testing

Exclusion Criteria:

* Currently participating in another research study
* Planning to move out of the Philadelphia area
* Unable to walk without pain
* Pregnant or planning to become pregnant in the year following study entry
* Excessive drinking
* Coronary heart disease
* Congestive heart failure
* Peripheral vascular disease
* Cerebrovascular disease
* Chronic obstructive pulmonary disease
* Arrhythmia
* Recurrent seizures
* Dizziness
* Balance problems
* Psychoses

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N. Sciamanna, MD, MPH, Study Chair — Jefferson Medical College, Department of Health Policy
Locations (2):
- United States (2):
  - Jefferson Family Medicine Associates, Philadelphia, Pennsylvania
  - Jefferson Medical College, Department of Health Policy, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Carroll JK, Lewis BA, Marcus BH, Lehman EB, Shaffer ML, Sciamanna CN. Computerized tailored physical activity reports. A randomized controlled trial. Am J Prev Med. 2010 Aug;39(2):148-56. doi: 10.1016/j.amepre.2010.04.005. PMID 20621262

RESULTS

PARTICIPANT FLOW:
Groups:
- Tailored Physical Activity Intervention Group: The intervention group completed physical activity surveys at baseline, 1, 3, and 6 months. Based on their responses, participants received four feedback reports at each time point. The reports aimed to motivate participants to increase physical activity, personalized to participants' needs; they also included an activity prescription.
- No Tailored Physical Activity Intervention Group: The control group received identical procedures, except that they received general reports on preventive screening based on their responses to preventive screening questions.
Period: Overall Study
Arm/Group | Tailored Physical Activity Intervention Group | No Tailored Physical Activity Intervention Group
Started | 187 | 207
Completed | 165 | 188
Not Completed | 22 | 19
Not completed — Lost to Follow-up | 22 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Physical Activity Intervention Group | No Tailored Physical Activity Intervention Group | Total
Number analyzed (Participants) | 187 | 207 | 394
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 187 | 207 | 394
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.2) | 48.4 (11.1) | 46.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 165 | 332
  Male | 20 | 42 | 62
Region of Enrollment [Number; unit: participants]
  United States | 187 | 207 | 394

OUTCOME MEASURES:

1. Primary Outcome: 7-Day Physical Activity Recall (7-Day PAR)
Description: Minutes of physical activity measured by the 7-Day Physical Activity Recall (7-Day PAR), which is an interviewer-administered self-report physical activity measure of minutes spent in moderate and vigorous intensity leisure and non-leisure activities over the preceding 7 days. It was administered to study participants at baseline and 6 months.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Tailored Physical Activity Intervention Group | No Tailored Physical Activity Intervention Group
Number analyzed (Participants) | 187 | 207
minutes | 54.85 [6.45 to 103.24] | 44.89 [3.19 to 86.59]

2. Secondary Outcome: Change in Behavioral Processes of Change Between Baseline and 6 Months
Description: Behavioral processes were assessed by asking participants to rate their responses to 24 statements on a Likert scale (1 = never to 5 = repeatedly) to statements such as, "I tell myself I am able to be physically active if I want to. To create the overall measure, individual items are averaged. Higher numbers represent greater use of behavioral processes of change, so that the overall scale retains a maximum of 5.0 and minimum value of 1.0. The scale values are not numerical, they represent scores on the scale, where 5=repeatedly and 1=never.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Tailored Physical Activity Intervention Group | No Tailored Physical Activity Intervention Group
Number analyzed (Participants) | 187 | 207
Scores on a Scale | 0.52 (0) [0.42 to 0.62] | 0.18 (0) [0.10 to 0.27]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were collected by participants contacting the research team. Serious and/or other non-serious adverse events were not collected/assessed.
Arm/Group | Tailored Physical Activity Intervention Group | No Tailored Physical Activity Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/187 | 0/207
Other Adverse Events (participants affected / at risk) | 0/187 | 0/207

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No